CLINICAL TRIAL: NCT01483404
Title: Identification of Microcirculation in Fracture of the Femural Neck: How Does the Intracapsular Hematoma Affect the Capillary Bloodflow in the Caput Femoris?
Brief Title: Identification of the Microcirculation of the Caput Femoris After Fracture of the Femoral Neck
Acronym: MicroFemNeck
Status: Withdrawn | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A10-30
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Microcirculation of the Caput Femoris
Keywords: microcirculation; caput femoris
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient with fracture of femural neck: All patient with fracture of the femural neck in the listed period of time
  Interventions: Procedure: Measurement with O2c

INTERVENTIONS:
Procedure: Measurement with O2c — Intra-surgery measurement of the microcirculation with the O2c device

SUMMARY:
This project investigates wether the intra-capsular hematoma, that often occurs after fracture of the femural neck, decreases the capillary blood flow of the caput femoris.

During operation the measuring device of the O2c-machine in placed on the joint capsula first and afterwards, after surgical opening of the capsula, on the femur directly. The integral of the microcirculation of both parts of the femur is measured in both settings. So the capillary blood flow is measured with the hematoma still in situ, eventually putting pressure on the caput femoris and after the capsula has been opened, the pressure relieved and the hematoma removed. Both measurements are compared for each patient.

The O2c-machine measures non-invasive with light waves and laser-doppler. The sounding rod is packed in a sterile tube to prevent any contamination of the operation site.

ELIGIBILITY:
Inclusion Criteria:

* medial fracture of the femural neck
* surgical treatment (hip replacement)

Exclusion Criteria:Polytrauma

* pathologic fracture
* conservative treatment
* soft tissue damage
* delay of surgery more than 3 days
* Immune default
* polytrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with fracture of the femural neck, who are treated in the University Hospital Aachen
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Microcirculation of the caput femoris befor the capsula of the joint is opend
  Four Values are measured:
  oxygen saturation local Hb local blood flow local blood velocity

SECONDARY OUTCOMES:
Microcirculaiton of the caput femoris after the capusla of the joint has been surgically opened and the hematoma has been removed
  Four values are measured:
  oxygen saturation local Hb local blood flow local blood velocity

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Pape, Univ-prof.MD, Study Chair — Chief of medicine
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany